CLINICAL TRIAL: NCT03380572
Title: Initial Experience With a New Laparoscopic Based Robotically Assisted Surgical System for Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Principal Investigator, Ravi Aggarwal, Clinical Research Fellow, Imperial College London
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SenhanceChole
Record Dates: First submitted 2017-12-11; First posted 2017-12-21 (Actual); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Biliary Colic; Cholecystitis
Keywords: Robotic Surgery
MeSH Terms: conditions — Cholecystitis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Senhance Cholecystectomy (Experimental): Cholecystectomy operation performed using Senhance robotic system
  Interventions: Device: Senhance Assisted Cholecystectomy
- Laparoscopic Cholecystectomy (Active Comparator): Cholecystectomy operation performed using standard laparoscopic instruments
  Interventions: Procedure: Laparoscopic Cholecystectomy

INTERVENTIONS:
Device: Senhance Assisted Cholecystectomy — Cholecystectomy performed using Senhance surgical robotic system
  Arms: Senhance Cholecystectomy
Procedure: Laparoscopic Cholecystectomy — Standard laparoscopic cholecystectomy
  Arms: Laparoscopic Cholecystectomy

SUMMARY:
The Senhance™ surgical robotic system, previously known as Telelap Alf-X (TransEnterix, Morrisville, NC, USA) has recently become available in the UK. It aims to provide the robotic benefits of greater accuracy, dexterity and control with similar operational costs to traditional laparoscopy.

Patients randomly received either a standard laparoscopic cholecystectomy or the Senhance assisted cholecystectomy based on scheduled surgery date. A prospectively maintained database of the first 20 patients undergoing cholecystectomy with the Senhance Surgical System was retrospectively interrogated and compared to a concurrently treated group of 20 laparoscopically treated patients during the same timeframe.

ELIGIBILITY:
Inclusion Criteria:

ASA I or II Confirmed diagnosis of biliary colic or cholecystitis Normal LFTs

Exclusion Criteria:

Patients unable tor unwilling to consent BMI >40

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Purkayastha, MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Senhance Cholecystectomy | Laparoscopic Cholecystectomy
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Senhance Cholecystectomy | Laparoscopic Cholecystectomy | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (13) | 48.4 (12.2) | 46 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 3 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Operative Time
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Senhance Cholecystectomy | Laparoscopic Cholecystectomy
Number analyzed (Participants) | 20 | 20
minutes | 86.5 [60.5 to 106.5] | 31.5 [26 to 41]

2. Secondary Outcome: Morbidity Data
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Senhance Cholecystectomy | Laparoscopic Cholecystectomy
Number analyzed (Participants) | 20 | 20
Participants | 3 | 5

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Senhance Cholecystectomy | Laparoscopic Cholecystectomy
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Senhance Cholecystectomy (N=20) | Laparoscopic Cholecystectomy (N=20)
Wound infection (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Bile leak (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/72/NCT03380572/Prot_SAP_001.pdf